CLINICAL TRIAL: NCT03906552
Title: Adiyaman University
Brief Title: Effects of Acupressure and Foot Massage on Pain During Heel Lancing in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Adiyaman University School of Health, Adiyaman University Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/1-5
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Acute Pain
Keywords: acupressure; massage; pain; neonate; heel lancing
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupressure group (Experimental): 2 neonates did not calm down before heel lancing; oxygen saturation and heart rate values of 2 neonates could not be monitored because the pulse oximeter tool probe was not fastened well.
  Acupressure was performed when the mother was holding the neonate on her arm. For two minutes, acupressure was performed in the acupressure points (Kun Lun (UB60) and Taixi (K3). Each point was applied acupressure for 60 seconds, and heel lancing was performed right after this procedure. The acupuncture points that Kun Lun (UB60) and Taixi (K3) are on the side of the ankle.
  Interventions: Other: nonpharmalogocial methods
- masssage group (Experimental): oxygen saturation and heart rate values of 2 neonates could not be monitored because the pulse oximeter tool probe was not fastened well; heel lancing could not be performed at the first attempt (2 neonates).
  Foot massage was performed when the mother was holding the neonate on her arm. Each neonate was given foot massage for two minutes, and heel lancing was performed right after the massage.
  Interventions: Other: nonpharmalogocial methods
- control group (No Intervention): oxygen saturation and heart rate values of 1 neonates could not be monitored because the pulse oximeter tool probe was not fastened well; heel lancing could not be performed at the first attempt (2 neonates).
  No application was made to theneonates in the control group before heel lancing procedure

INTERVENTIONS:
Other: nonpharmalogocial methods — neonates received acupressure (acupressure group) or massage (massage group) before heel lancing procedure
  Arms: acupressure group; masssage group

SUMMARY:
Aim: The study was aimed to identifying the effects of foot massage and acupressure on pain during heel lancing in neonates.

Methods: A single-blinded randomized controlled trial was performed in a university hospital in Turkey between April-December 2018. Neonates were randomized into three groups as acupressure, massage and control groups. Data were obtained by using Information form, Neonatal Infant Pain Scale (NIPS), pulse oximeter device and chronometer. Acupressure was applied to the neonates in the acupressure group and massage was given to the neonates in the massage group for 2 minutes before heel lancing procedure. Pain levels of the neonates in the groups were evaluated during and 1 minute after heel lancing procedure. Furthermore, the oxygen saturation and heart rate values of the neonates in the groups were measured by pulse oximeter device before, during and after heel lancing procedure. Duration of crying and heel lancing procedure were recorded by chronometer.

DETAILED DESCRIPTION:
Massage is a systematic and scientific procedure applied by using hands or special tools. As for acupressure, it is a method applied by stimulating the acupuncture points using hands and fingers by applying pressure on the meridians in body.Both methods are reliable, economic and easy to learn and apply. Review of the related literature indicates studies on the effectiveness of acupressure and foot massage on reducing pain in neonates.

ELIGIBILITY:
Inclusion Criteria:

* having 2500-4000 gr body weight and being term neonates,
* having APGAR score of over 7 five minutes after birth,
* having no health problems detected in the newborn examination after birth,
* having received no painful interventions apart from Hepatitis B and Kvit after birth,
* being with the mother and being fed orally,
* having had breast milk within 30 minutes before heel lancing
* having a clean diaper.

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pain Scale | 1 minute
  Neonatal Infant Pain Scale (NIPS): The scale was developed by Lawrence et al. in 1993 in order to asses the behavioral and physiological pain responses of premature and term neonates. The scale consists of five behavioral and one physiological sections including facial expression, crying, breathing, arm and leg movements, and alertness. Total scores range between 0 and 7. Scores from 0 to 2 indicate mild to no pain, 3 to 4 indicates mild to moderate pain, and >4 indicates severe pain. Higher scores indicate more severe pain. In the study of Lawrence et al., NIPS 's Cronbach's Alpha 0.92 found (Larwence et al. 1993). The scale was adapted to Turkish by Akdovan, NIPS is used for the assessment of procedural pain of the premature and term neonates. Akdovan found the Cronbach's Alpha value to be 0.83. The pain intensity of neonates was evaluated during and 1 minute after heel lancing procedure

OTHER OUTCOMES:
Pulse Oximeter Device | 1 minute
  It was used for the measurement of oxygen saturation and heart rate before, during and after heel lancing in all three groups.
Chronometer | 2 minutes
  Duration of crying and heel lancing procedure were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Adiyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided